CLINICAL TRIAL: NCT02569489
Title: Phase I Dose Escalation Study of HBI-8000 in Combination With Paclitaxel and Trastuzumab in Women With Advanced or Metastatic HER2+ Breast Cancer
Brief Title: Dose Escalation Study of HBI-8000 in Combination With Paclitaxel and Trastuzumab in Women With Advanced or Metastatic HER2+ Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Reconsideration of Study Design; plan for alternative protocol
Sponsor: HUYABIO International, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI-8000-106
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2016-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — HBI-8000; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HBI-8000, Paclitaxel, Trastuzumab (Experimental): HBI-8000 at the assigned dose twice weekly while receiving weekly paclitaxel and trastuzumab for a minimum of 8 weeks (2 treatment cycles)
  Interventions: Drug: HBI-8000; Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: HBI-8000
Drug: Trastuzumab
Drug: Paclitaxel

SUMMARY:
This is a phase I multi-center dose escalation study of the histone deacetylase inhibitor (HDACi) HBI-8000 when given in combination with paclitaxel and trastuzumab in women with advanced or metastatic HER2+ breast cancer.

DETAILED DESCRIPTION:
This is a phase I multi-center dose escalation study of the histone deacetylase inhibitor (HDACi) HBI-8000 when given in combination with paclitaxel and trastuzumab in women with advanced or metastatic HER2+ breast cancer.

Three dose levels of HBI-8000 (15 mg, 20 mg, and 25 mg) will be tested using a standard 3+3 escalation plan with an expanded cohort at the maximum tolerated dose (MTD) to enroll a minimum of 10 patients evaluable for safety to fulfill the requirements for moving the combination forward to I-SPY 2 trial.

To be considered evaluable for safety, the patient must receive at least 75% of their prescribed regimen per cycle for 4 consecutive cycles with a cycle of therapy defined as 28 days in the absence of disease progression or unacceptable toxicity. Patients who progress at 9 weeks evaluation or later but before completing 4 cycles and who have only experienced Grade ≤ 1 toxicities (excluding alopecia) will also be considered evaluable for safety.

Enrolled patients will remain on their assigned dose level until unacceptable toxicity or disease progression occurs. During dose escalation phase, if more than 34% of the evaluable patients at a dose level experience dose limiting toxicities (DLT), this dose level will be considered having exceeded MTD. Once MTD is identified during dose escalation phase, the MTD dose level will be expanded in the expansion phase to enroll additional patients to ensure that at least 10 patients are evaluable for safety at the MTD.

Paclitaxel and trastuzumab are administered by intravenous (IV) infusion on days 1, 8, 15, and 22 of a 28-day cycle. HBI-8000 will be taken by mouth twice weekly at the assigned dose on days 1, 4, 8, 11, 15, 18, 22 and 25 of a 28-day cycle. Treatment continues until disease progression, unacceptable toxicity, or patient refusal/non-compliance is observed.

The study will evaluate the safety and tolerability of oral HBI-8000 bi-weekly in combination with weekly paclitaxel and trastuzumab and if successful, determine an optimal dose to move into phase II testing of this combination in the I-SPY 2 trial in a neo-adjuvant breast cancer population.

To determine the MTD of HBI-8000 twice weekly in combination with weekly paclitaxel and trastuzumab in women with HER2+ breast cancer.

* To determine the adverse event rate of twice weekly HBI-8000 in combination with weekly paclitaxel and trastuzumab
* To determine the tolerability of twice weekly HBI-8000 when administered with weekly paclitaxel and trastuzumab
* To explore efficacy of twice weekly HBI-8000 in combination with weekly paclitaxel and trastuzumab
* To obtain pharmacokinetics of twice weekly HBI-8000 when administered in combination with weekly paclitaxel and trastuzumab.
* To determine the on-target effect of HBI-8000 by measuring protein acetylation
* To explore the treatment effects on immune cells in blood and/or tumor tissue as appropriate

Enrolled patients will take HBI-8000 at the assigned dose twice weekly while receiving weekly paclitaxel and trastuzumab for a minimum of 8 weeks (2 treatment cycles). On the day of paclitaxel infusion, HBI-8000 is taken at least one hour before paclitaxel infusion. HBI-8000 should be taken within 30 minutes after a meal. The interval between HBI-8000 administrations is 3-4 days in the absence of dose delay or interruptions due to adverse events. For example, three days should elapse between the 1st and 2nd dose of HBI-8000 of the week, such as Monday/Thursday; Tuesday/Friday.

A disease re-evaluation will be scheduled every 8 weeks. Based on the Response Evaluation Criteria in Solid Tumors 1.1 (RECIST1.1), response to treatment will be determined. Patients with stable disease (SD), partial response (PR) or complete response (CR) may continue treatment until disease progression, unacceptable side effects, or patient refusal/non-compliance occurs.

Patients will be monitored in clinic every 4 weeks while receiving study treatment. The end of treatment (EOT) visit will occur at 4 weeks after the last dose of HBI-8000, or before the start of a new anti-cancer therapy, whichever is earlier. At EOT, patients will be evaluated for resolution of treatment related toxicities. Toxicity related to HBI-8000, if not yet resolved to Grade ≤ 1, will be followed until resolution to Grade ≤ 1 or considered chronic. All patients will be followed up to 1 year from study enrollment for best objective response, duration of response, time to PD, and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Female subject, age ≥18 years at the time of signing informed consent
2. Histologically or cytologically confirmed adenocarcinoma of breast, HER2+ as determined by FISH or IHC
3. Having received at least one prior systemic therapy with FDA approved agent(s) for metastatic disease and have no curative option
4. Measureable disease as defined by RECIST 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
6. Laboratory parameters within 14 days prior to dosing:

   * Absolute neutrophil count (ANC) ≥ 1.5 X 109/L independent of growth factor support
   * Hemoglobin (Hgb) ≥9 gm/dL independent of transfusion or growth factor support
   * Platelets (plt) ≥ 100 x 109/L independent of transfusion or growth factor support
   * AST and ALT ≤2.5 x Upper Limit of Normal (ULN); if hepatic metastasis is present, ≤2.5 x ULN
   * Serum total bilirubin ≤ 1.5 x ULN; if with Gilbert's Syndrome, direct bilirubin must be normal
   * Serum creatinine ≤ 1.5 x ULN or eGFR ≥ 60ml/min
   * Serum albumin > 3.0 g/dL
   * Prothrombin time (PT)/International normalized ratio (INR) ≤ 1.5, partial thromboplastin time (PTT) within normal limits (WNL) of the institution
7. Negative serum pregnancy test in subjects with child-bearing potential; and commit to abstinence or comply with medically proven contraception methods
8. Agree to abstain from breast feeding from the start of study treatment and >28 days after the last dose of study drugs.
9. Understand and voluntarily sign informed consent

Exclusion Criteria:

1. Receiving chemotherapy, immunotherapy, biological, radiation therapy or investigational agent (therapeutic or diagnostic) within 4 weeks prior to receipt of study medication. Major surgery, other than diagnostic surgery, within 4 weeks before first study drug administration.
2. Significant cardiac history:

   * History of myocardial infarction or ischemic heart disease within 1 year before the first study drug administration
   * Uncontrolled arrhythmia, such as ventricular tachycardia, ventricular fibrillation; second- or third-degree heart block; unstable angina, coronary angioplasty or stenting, or myocardial infarction (MI) within 6 months of study entry
   * History of congenital QT prolongation, or baseline QTcF > 470 ms using Fridericia's formula
   * ECG findings consistent with active ischemic heart disease
   * New York Heart Association Class III or IV cardiac disease
   * Left ventricular Ejection Fraction measuring ≥ 55% at baseline ECHO
   * Uncontrolled hypertension: blood pressure consistently greater than 150 mm Hg systolic and 100 mm Hg diastolic in spite of antihypertensive medication
3. Patients with active brain metastasis or leptomeningeal involvement. Patients who have brain metastases that have been previously treated, who are asymptomatic, and whose lesions by imaging are at least stable and without interim development of new lesions for at least 6 weeks may be enrolled. Patients who require continued steroid therapy as management for their brain metastases are not eligible
4. Persistent diarrhea or malabsorption NCI CTCAE (version 4.03) grade ≥ 1 despite medical management, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting GI function
5. Peripheral neuropathy NCI CTCAE (Version 4.03) Grade ≥ 2
6. Active uncontrolled bacterial, viral, or fungal infection requiring systemic therapy.
7. Known infection with human immunodeficiency virus (HIV) or active hepatitis A, B, or C.
8. Patients with a prior hypersensitivity reaction to any product containing polyvinylpyrrolidone, microcrystalline cellulose, lactose monohydrate, sodium starch glycolate, talc or magnesium stearate.
9. Second malignancy unless in remission for > 5 years. (Non-melanoma skin cancer or carcinoma in situ of the cervix treated with curative intent is not exclusionary.)
10. Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient. Examples of such conditions include infection requiring parenteral anti-infective treatment, hydronephrosis, liver failure, any altered mental status or any psychiatric condition that would interfere with the understanding of the informed consent.
11. Unwilling or unable to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Estimated); Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
MTD of HBI-8000 twice weekly in combination with weekly paclitaxel and trastuzumab in women with HER2+ breast cancer | 28 days